CLINICAL TRIAL: NCT06478836
Title: Does Planter Pressure and Body Mass Index Affect Balance in Normal Children
Brief Title: Planter Pressure and Body Mass Index Affect Balance in Normal Children
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa S Ali, associate professor of pediatric physiotherapy, cairo university, Cairo University
Other Study IDs: P.T.REC/012/ 004586
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Plantar Pressure
Keywords: association; foot pressure; body mass index; balance; normal children

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: planter pressure — no intervention

SUMMARY:
is there relation between planter pressure, body mass index and balance in normal children?

DETAILED DESCRIPTION:
is there relation between planter pressure, body mass index and balance in normal children?

ELIGIBILITY:
Inclusion Criteria:

* Normal children from both sex
* Age from 8 to 12 years

Exclusion Criteria:

* recent fractures or procedures
* open wounds on the lower limbs,
* any fixed deformities in the lower limbs

Ages: 8 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: One hundred normal children aged from 8 to 12 years old will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-07-23 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Foot pressure will be recorded by a pedograph | 3 months
  Foot pressure will be recorded by a pedograph
BMI will be calculated by weight/height^2 (CDC chart). | 3 months
  BMI will be calculated by weight/height^2 (CDC chart).
Balance will be assessed by Biodex | 3 months
  Balance will be assessed by Biodex

CONTACTS AND LOCATIONS:
Locations (1):
- Mostafa S Ali, Giza, Married, Egypt

REFERENCES:
- [Derived] Ali MS, Aly SM, Usama M. Relationship Between Plantar Pressure, Body Mass Index and Balance in Children: A Cross-Sectional Study. J Musculoskelet Neuronal Interact. 2025 Dec 1;25(4):414-421. doi: 10.22540/JMNI-25-414. PMID 41324212